CLINICAL TRIAL: NCT06567184
Title: Pilot Evaluation of the Strong Hearts Program in an Urban Setting
Brief Title: Evaluation of the Strong Hearts Urban Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB2022-0801D
Record Dates: First submitted 2024-08-14; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Strong Hearts Urban (Experimental): A 12-week multi-level intervention targeting behavior modification, nutrition education, strength training, aerobic exercise, and stress reduction activities
  Interventions: Behavioral: Strong Hearts Urban

INTERVENTIONS:
Behavioral: Strong Hearts Urban — A 12-week multi-level intervention targeting behavior modification, nutrition education, strength training, aerobic exercise, and stress reduction activities

SUMMARY:
The aim of this study is to assess the feasibility and preliminary effectiveness of the adapted Strong Hearts (SH) intervention to improve weight status, American Heart Association's Life's Essential 8 (AHA Essential 8), and health behaviors among Black/African American and/or Hispanic/Latinx urban residents with overweight or obesity.

DETAILED DESCRIPTION:
Cultural adaptation of effective health behavior interventions holds the potential to improve health behaviors and ultimately health outcomes among underserved populations. The Strong Hearts (SH) Urban Intervention will adapt the existing SH curriculum for delivery in urban Dallas communities to improve weight status and Life's Essential 8 score for ideal cardiovascular health. Despite declines in heart disease mortality in the United States since 2000, it remains the leading cause of mortality in both men and women-accounting for about one-third of all deaths in the U.S. Costs related to cardiovascular disease (CVD) place a substantial financial burden on the health care system, accounting for an estimated $320 billion in 2016. Although most obesity or CVD prevention programs target only the individual level, the US Centers for Disease Control and Prevention recognizes that health is affected by factors at multiple levels: individual (e.g., behaviors, knowledge, attitudes, skills, psychological factors), social (e.g., influences from one's social network on health-related behaviors), and environmental (e.g., safe places to walk, food choices at workplaces, availability of affordable fruits and vegetables), and recommends integrating approaches to make changes beyond the individual level to support long-term, sustainable behavior change. Providing individuals with the motivation, skills, and opportunity to change behaviors may be less effective if their social or community environment makes it difficult to adopt or maintain these behaviors

SH is a multilevel, multicomponent community-based program, in which an experiential learning focus is combined with social and environmental components, including civic engagement activities related to local resource awareness and enhancement. There is limited knowledge about how programs and services can move beyond commonly used individual-level approaches, which have limitations in terms of cost, impact, reach, and sustainability, to effectively reduce CVD health disparities using an integrated, multi-level, community-engaged approach. This pilot study will provide needed data on the feasibility and preliminary effectiveness of such approaches in urban and underserved communities.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 or older
2. Overweight or obese (BMI≥25)
3. Less than 150 minutes of moderate physical activity per week
4. Black/African American race and/or Hispanic/Latinx ethnicity

Exclusion Criteria:

1. Pregnancy, or intent to become pregnant during the study duration
2. Unable to read and communicate in English
3. Planning to participate in another health behavior change program in the next three months
4. Unable/unwilling to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — What is your gender?
Enrollment: 51 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Body Weight | 12 weeks
  Change in body weight

SECONDARY OUTCOMES:
Fruit and Vegetable Consumption | 12 weeks
  Dermal Carotenoid Score. As measured by Veggie Meter using a participant's index finger, the dermal carotenoid score (0-800) reflects a concentration biomarker of fruit and vegetable intake, where a higher score is correlated with higher intake.
Self-reported healthy eating behaviors | 12 weeks
  Healthy Eating Index (HEI) as measured by Dietary Health Questionnaire (DHQ-III). The DHQ-III is a self-administered, web-based food frequency questionnaire scored 0 to 100, where higher scores indicate closer adherence to the Dietary Guidelines for Americans.
Physical activity - Active Minutes | 12 weeks
  Objectively measured physical activity by Fitbit activity tracker, counted as Active Minutes
Physical activity - Steps | 12 weeks
  Objectively measured physical activity by Fitbit activity tracker, counted as steps
Participant Acceptability | 12 weeks
  Participant feedback from follow-up questionnaires measures acceptability on a 5-point Likert scale, where higher score indicates higher satisfaction
Intervention Engagement | 12 weeks
  Engagement is assessed by attendance at study activities including intervention classes and data collection appointments

CONTACTS AND LOCATIONS:
Overall Officials: Chad D Rethorst, Ph.D., Principal Investigator — Texas A&M AgriLife Research
Locations (2):
- United States (2):
  - West Dallas Multipurpose Center, Dallas, Texas
  - Texas A&M AgriLife Research and Extension Center at Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No